CLINICAL TRIAL: NCT02378298
Title: Rituximab (RTX) Therapy in Steroid Resistant Patients or Patients Relapsing After Intravenous Steroids With Active TAO
Brief Title: Rituximab (RTX) Therapy in Patients With Active TAO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RTX -TAO
Record Dates: First submitted 2015-01-20; First posted 2015-03-04 (Estimated); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Ophthalmopathy, Thyroid-Associated
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Rituximab; Methylprednisolone; Methylprednisolone Hemisuccinate; Methotrexate; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Non-responder RTX+MTX (Active Comparator): Patients with moderate-severe TAO with an inflammatory CAS of ≥ 4 that do not respond to iv GC (deltaCAS <2 compared to baseline after 4 weeks of iv GC ) or do relapse (deltaCAS ≥2 and total CAS ≥4) after steroid treatment compared to previous CAS measurement at 12 weeks. Rituximab (1000 mg iv with 2 weeks in between) is combined with methotrexate (15-20 mg once a week) to minimize the risk of antibody developement. MTX is always combined with RTX and is never given as a monotherapy in this study.
  rituximab and methotrexate
  Interventions: Drug: Rituximab
- Relapse RTX+MTX (Active Comparator): Patients that respond to iv GC (Methylprednisolone iv) but relapse after 6 weeks will be randomised to either RTX+MTX or per oral GC (po GC+MTX) rituximab and methotrexate
  Interventions: Drug: Rituximab
- Relapse po GC+MTX (Active Comparator): Patients that respond to iv GC but relapse after 6 weeks will be randomised to either RTX+MTX or per oral GC (po GC+MTX) This is the conventional therapy arm.
  methotrexate and methylprednisolone
  Interventions: Drug: peroral methylprednisolone and Methotrexate
- Responders without relapse (No Intervention): Patients that respond to iv GC and have no relapse at 18 weeks of study.
- Methylprednisolone iv (Active Comparator): All patients in the study have a 4 weeks period of 500 mg methylprednisolone iv/week. Depending of the response patients are classified as non- responders (and are given RTX and MTX) or responders. The responders continue with intravenous infusion of Methylprednisolone 500 mg /week in 2 weeks and thereafter 250 mg iv/week in 6 weeks.
  Interventions: Drug: Iv Methylprednisolone

INTERVENTIONS:
Drug: Rituximab — Rituximab (RTX) is a mouse-human chimeric antibody designed towards (CD20) pre B and mature B lymphocytes and that blocks B-cells activation without affecting the regenerating of B cells from stem cells or the plasma cells immunoglobulin production. Rituximab is used in the treatment of hematologic malignancies (B cells lymphoma, chronic lymphatic leukaemia, Waldenströms macroglobulinemia) and autoimmune diseases with B-cell involvement such as rheumatoid arthritis, thrombocytopenic purpura, SLE).
  Other Names: Mabthera; Rituxan; Zytux; L01XC02
  Arms: Non-responder RTX+MTX; Relapse RTX+MTX
Drug: Iv Methylprednisolone — Solumedrol is an intravenous glucocorticoid that are the gold standard in TAO. All patients start with 500 mg/weeks for 4 weeks. The response is evaluated and patients are randomised to non-responders or responders. The responders continues with the gold standard treatment that is another 500 mg solumedrol/ week in 2 weeks and then 250 mg/ week in 6 weeks.
  Other Names: Solumedrol
  Arms: Methylprednisolone iv
Drug: peroral methylprednisolone and Methotrexate — Peroral GC (starting with 30 mg and tapering down) is combined with 15-20 mg MTX /week to reduce the needed dose of steroids
  Other Names: Prednisolone
  Arms: Relapse po GC+MTX

SUMMARY:
Thyroid Associated Ophthalmopathy is condition affecting the eyes of about 10% of patients with Graves disease. Its combination of protrusion affecting the looks of the patient and pain is often severely affecting the quality of life among these patients.

The standard treatment for this illness today is intravenous glucocorticoids together with methotrexate. The purpose of this study is to evaluate the effect of rituximab on patients that do not respond to or relapse after conventional therapy.

DETAILED DESCRIPTION:
Diffuse autoimmune hyperthyroidism or Graves' disease (GD) is a common condition mainly affecting women with 2-3% prevalence The increased production of thyroid hormones in GD is driven by autoantibodies directed against the thyroid stimulating hormone (TSH) receptor (TRab). In most cases, this autoimmunity will also affect other tissues, above all the orbital tissue by mechanisms not fully understood -Thyroid Associate Ophthalmopathy (TAO). Symptoms and signs can be mild (grittiness, dry eyes, periorbital swollen, chemosis, redness)-moderate (double eye vision, exophthalmia or severe (optic nerve compression, corneal ulcers). Serious-moderate ocular engagement in TAO is seen in approximately 10% of patients with GD.

Not only has the hyperthyroidism a marked impact on mental health, but the presence of TAO has an additional negative impact on the well-being of these patients, even many years after successful treatment of the hyperthyroidism. It has been suggested that smoking and stress are negative prognostic factors for the course of TAO indicating that a vicious circle. MRI may detect earlier changes than CT that can be used to predict the course of TAO.

The aims of treatment are to retain euthyroidism which can be achieved by anti thyrostatic drugs (ATD), radioiodine treatment or surgery (where patients are pre-treated with ATD) and to avoid TAO as long as possible. If moderate-severe TAO occurs, high dose if intravenous glucocorticoids (GC) are the gold standard considering the side effects. However, many patients are non-steroid responders and for them no treatment except for acute orbital decompression, retro bulbar irradiation and later reconstructive surgery can be offered. When patients relapse immediately after steroids often per oral steroids are given although not recommended from the literature.

Rituximab (RTX) is a mouse-human chimeric antibody designed towards pre B and mature B lymphocytes and that blocks B-cells activation without affecting the regenerating of B cells from stem cells or the plasma cells immunoglobulin production. TAO is a B- lymphocyte mediated disease and in two studies RTX inhibits the active phase of TAO. In a study by Khanna et al a positive effect from RTX is observed in six steroid resistant patients with TAO with a decrease of the inflammation in the orbit, even though no effect on strabismus or proptosis was observed. In another study by Salvi et al , RTX treatment is compared with steroids as a first line treatment for TAO and after 30 weeks of follow up in an unrandomised study design. RTX decreased the activity and severity significantly compared to the steroid group. No relapse was observed in the RTX group but in the steroid group (10%). In the RTX all patients improved, but in the steroid group only 65%. There were more side-effects in the steroid group.

Selection criteria All patients with indication for i.v GC will be evaluate for the study. The patients are recruited consecutively from the region as we are a tertial referral center and iv steroids for TAO is not given on local hospitals..

Patients and study design All patients aged 18-70 years in the western region in Sweden with TAO and indication for iv GC (CAS ≥4) will be evaluated for this prospective open study with RTX+MTX to GC non-responders. If GC respondent but relapsing after 12 weeks of iv GC treatment, patients will be randomized to RTX+MTX or per oral GC+MTX. If non respondent after 4 weeks of intravenous steroid infusion the patient will be eligible for RTX treatment Patients are seen for ophthalmological and endocrine investigations at baseline, 4, 12, 18, 32, 44, 56 and 68 weeks. At similar occasions anthropometric measurements, immunological markers and measures of GC effects (ACTH test, body composition (not all occasions)) will be performed. At baseline and after 30 weeks high quality MRI and Gallium (GA)-PET is performed. Patients undergoing Ga-PET in another study focusing on pituitary imaging (principle investigator HFN) will serve as controls for orbital muscles. The aim of the RTX study is to recruit at least 10 patients in the RTX arm and probably 40-50 patients will be included.

No study with this design has previously been published. The present situation does not offer the patients not responding to GC or with relapses after iv GC infusions any effective treatment. If the RTX proves safe and effective future non-respondent patients will be able to get this treatment. In small studies RTX have had a good effect in TAO, sometimes even better than GC and with less side-effects. It will also lay the ground for future studies that compare RTX and GC in a randomised study design as first line treatment. If GA-PET shows useful in the management of patients with TAO it may become a routine investigation.

ELIGIBILITY:
Inclusion Criteria:

* ◦Man or woman between 18-70 years TAO with CAS of ≥ 4 (less than 3 months).
* Euthyroid for at least 6 weeks

Exclusion Criteria:

* Dysthyroid optic neuropathy (DON)
* Ulcerative Keratitis
* Previous treatment with steroids for TAO (do not include prophylaxis for TAO in connection with radio iodine treatment)
* Previous Treatment with Rituximab (MabThera®)
* Positive Hepatitis B or C serology.
* Receipt of a live vaccine within 4 weeks prior RTX+MTX to randomization
* History of recurrent significant infection or history of recurrent bacterial infections
* Patient who may not attend to the protocol according to the investigators opinion.
* Pregnancy or lactation
* Significant cardiac, including significant or uncontrolled arrhythmia, or pulmonary disease (including obstructive pulmonary disease).
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Concomitant malignancies or previous malignancies.
* Previous active tuberculosis
* Alcoholism
* Alcoholic related liver disease or other chronical liver disease
* Bone marrow depression with leukopenia, thrombocytopenia or significant anemia
* Rheumatoid or other significant pulmonary disease
* Allergy to the active substance or any other substance in the medications or murine proteins
* Active, severe infections (such as tuberculosis, sepsis or opportunistic infections)
* Patients with severe immunosuppression
* Severe cardiac failure or severe uncontrolled heart disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Filipsson, Ass Prof, Principal Investigator — Sahlgrenska University Hospital
Locations (5):
- Sweden (5):
  - Center for Endocrinology and Metabolism, Sahlgrenska University Hospital, Gothenburg
  - MedTech West, Institute of Neuro Science and Physiology, Department for Clinical Neuro Science and Rehabilitation, Sahlgrenska Academy, University of Gothenburg, Gothenburg
  - Department of Ophthalmology, Sahlgrenska University Hospital/Mölndal, Mölndal
  - Department of Rheumatology, Sahlgrenska University Hospital/Mölndal, Mölndal
  - Department of Radiology, Karolinska University Hospital, Stockholm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Enrollment number in the Protocol Section (38) conflicts with the number of participants Started in the Participant Flow module (37). The allocation to the groups (NR-RTX or R-GC) depends on the assessment of the participants' response AT 4 WEEKS. Since one participant dropped-out during the run-in period, i.e. BEFORE the evaluation at 4 weeks, this participant was NOT assigned to an Arm/Group during the Run-In period and can therefore not be included in results reported in a tabular format.
Groups:
- Responders (R-CG): All patients in the study have a 4 weeks period of 500 mg methylprednisolone iv/week. Depending of the response patients are classified as non- responders (and are given RTX and MTX) or responders. The responders continue with intravenous infusion of Methylprednisolone 500 mg /week in 2 weeks and thereafter 250 mg iv/week in 6 weeks.
- Non-responders RTX+MTX (NR-RTX): Patients with moderate-severe TAO with an inflammatory CAS of ≥ 4 that do not respond to iv GC (deltaCAS <2 compared to baseline after 4 weeks of iv GC ) or do relapse (deltaCAS ≥2 and total CAS ≥4) after steroid treatment compared to previous CAS measurement at 12 weeks. Rituximab (1000 mg iv with 2 weeks in between) is combined with methotrexate (15-20 mg once a week) to minimize the risk of antibody developement. MTX is always combined with RTX and is never given as a monotherapy in this study.
  rituximab and methotrexate
- Non-responders Control Group (R-C): A retrospective group of non-responsive patients after 4 weeks with iv glucocorticoids, who received regular care, i.e. full 12-week treatment with glucocorticoids according to clinical praxis. This group was used as control and received the same therapy as Responders (R-CG).
Period: Run-In (0-4 Weeks)
Arm/Group | Responders (R-CG) | Non-responders RTX+MTX (NR-RTX) | Non-responders Control Group (R-C)
Started | 13 | 12 | 12
Completed | 13 | 10 | 12
Not Completed | 0 | 2 | 0
Not completed — development of dysthyroid optic neuropathy | 0 | 2 | 0
Period: Intervention (5-12 Weeks)
Arm/Group | Responders (R-CG) | Non-responders RTX+MTX (NR-RTX) | Non-responders Control Group (R-C)
Started | 13 | 10 | 12
Completed | 13 | 10 | 11
Not Completed | 0 | 0 | 1
Not completed — As a deviation from the clinical praxis, withdrew the subject from the regular therapy | 0 | 0 | 1
Period: Follow-up (13-18 Weeks)
Arm/Group | Responders (R-CG) | Non-responders RTX+MTX (NR-RTX) | Non-responders Control Group (R-C)
Started | 13 | 10 | 11
Completed | 13 | 10 | 11
Not Completed | 0 | 0 | 0
Period: Surveillance (19-68 Weeks)
Arm/Group | Responders (R-CG) | Non-responders RTX+MTX (NR-RTX) | Non-responders Control Group (R-C)
Started | 13 | 10 | 11
Completed | 12 | 10 | 11
Not Completed | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-responders RTX+MTX (NR-RTX) | Responders (R-CG) | Non-responders Control Group (R-C) | Total
Number analyzed (Participants) | 12 | 13 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (9.1) | 54.6 (6.9) | 57.5 (12.0) | 55 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 7 | 25
  Male | 6 | 1 | 5 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Smoking status [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    Smoker | 7 | 2 | 5 | 14
    Previous smoker | 4 | 9 | 2 | 15
    Non-smoker | 1 | 2 | 3 | 6
    Unknown | 0 | 0 | 2 | 2
Thyroid-stimulating hormone receptor antibodies [Median (Inter-Quartile Range); unit: International Units per Liter] — Thyroid-stimulating hormone receptor antibodies (TRAb) Population: Blood sample missing.
  International Units per Liter
    number analyzed (Participants) | 11 | 11 | 11 | 33
    (all) | 28.6 [7.8 to 41.0] | 11.4 [5.9 to 20.3] | 9.7 [4.7 to 27.0] | 11.4 [5.7 to 29.5]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Activity Score (a Composite Measure of Ophthalmological Signs and Symptoms)
Description: Clinical activity score (CAS) according to Mouritz et al and the consensus statement from European Group of Graves orbitopathy (EUGOGO). It consists of 10 items (1. Spontaneous retrobulbar pain, 2. Pain on eye movements, 3. Eyelid erythema, 4. Conjunctival injection, 5. Chemosis, 6. Swelling of the caruncle, 7. Eyelid edema or fullness, 8. Change in motility,9. Change in vision acuity,10.Change in proptosis). One point is given to each item, if present. CAS is the sum of single scores, ranging from 0 (no activity) to 10 (maximal activity).
Time Frame: At 4,12,18 and 68 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-responders RTX+MTX (NR-RTX) | Responders (R-CG) | Non-responders Control Group (R-C)
Number analyzed (Participants) | 12 | 13 | 12
score on a scale
  at 4 weeks | 4.25 (0.99) | 2.77 (1.36) | 4.25 (0.87)
  at 12 weeks | 4.20 (1.03) | 2.88 (1.33) | 4.00 (1.41)
  at 18 weeks | 4.05 (1.23) | 3.81 (1.35) | 3.63 (1.60)
  at 68 weeks | 3.00 (1.39) | 2.58 (1.40) | 2.14 (2.12)

2. Other Pre Specified Outcome: Thyroid-stimulating Hormone Receptor Antibodies
Time Frame: at 4 weeks
Measure: Median (Inter-Quartile Range); unit: International Units per Liter
Arm/Group | Non-responders RTX+MTX (NR-RTX) | Responders (R-CG) | Non-responders Control Group (R-C)
Number analyzed (Participants) | 10 | 13 | 5
International Units per Liter | 23.5 [3.6 to 41.0] | 7.7 [2.6 to 12.5] | 3.9 [1.7 to 10.1]

3. Other Pre Specified Outcome: Thyroid-stimulating Hormone Receptor Antibodies
Time Frame: at12 weeks
Measure: Median (Inter-Quartile Range); unit: International Units per Liter
Arm/Group | Non-responders RTX+MTX (NR-RTX) | Responders (R-CG) | Non-responders Control Group (R-C)
Number analyzed (Participants) | 10 | 12 | 10
International Units per Liter | 15.0 [1.8 to 32.8] | 2.1 [0.8 to 4.4] | 8.1 [1.5 to 20.7]

4. Other Pre Specified Outcome: Thyroid-stimulating Hormone Receptor Antibodies
Time Frame: at18 weeks
Measure: Median (Inter-Quartile Range); unit: International Units per Liter
Arm/Group | Non-responders RTX+MTX (NR-RTX) | Responders (R-CG) | Non-responders Control Group (R-C)
Number analyzed (Participants) | 10 | 13 | 4
International Units per Liter | 11.9 [1.5 to 32.0] | 3.8 [0.9 to 5.0] | 1.6 [0.7 to 8.1]

5. Other Pre Specified Outcome: Thyroid-stimulating Hormone Receptor Antibodies
Time Frame: at 68 weeks
Measure: Median (Inter-Quartile Range); unit: International Units per Liter
Arm/Group | Non-responders RTX+MTX (NR-RTX) | Responders (R-CG) | Non-responders Control Group (R-C)
Number analyzed (Participants) | 9 | 9 | 5
International Units per Liter | 1.9 [0.7 to 22.0] | 2.1 [0.7 to 11.0] | 4.0 [0.7 to 9.1]

ADVERSE EVENTS:
Time Frame: Intervention phase = 4-12 weeks Follow-up phase: 13-18 weeks Surveillance phase: 19-68 weeks
Description: Data on Adverse events was collected only for the R-GC and NR-RTX during the 3 phases: intervention, follow-up & surveillance. Data on adverse events was NOT collected during the run-in phase, ie. prior to start of the tested intervention Rituximab. During the run-in phase the participants received regular care according to clinical praxis. Data on adverse events was NOT collected from the NR-RC group, as the data related to this control group was collected retrospectively from medical journal.
Arm/Group | Non-responders RTX+MTX (NR-RTX) | Responders (R-CG)
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/13
Serious Adverse Events (participants affected / at risk) | 2/10 | 0/13
Other Adverse Events (participants affected / at risk) | 8/10 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-responders RTX+MTX (NR-RTX) (N=10) | Responders (R-CG) (N=13)
Mental disorder (Nervous system disorders) | 1 (1) | 0 (0) — Inpatient care due to mental disorder
Cerebral aneurysm (Nervous system disorders) | 1 (2) | 0 (0) — Inpatient care when cerebral aneurysm was diagnosed and new event of inpatient care for operation of aneurysm in the same individual
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-responders RTX+MTX (NR-RTX) (N=10) | Responders (R-CG) (N=13)
High blood pressure (Cardiac disorders) | 5 (7) | 7 (11) — Systolic blood pressure > 140 or diastolic blood pressure > 90
High liver tests (Hepatobiliary disorders) | 0 (0) | 1 (1) — 3-fold elevation of AST or ALT
Positive oral glucose tolerance test (Endocrine disorders) | 3 (4) | 2 (4) — Diabetes or glucose intolerance
Inadequate response to short ACTH (Endocrine disorders) | 0 (0) | 1 (1) — A short ACTH test was conducted by measuring serum cortisol at 0, 30, and 60 min after IV ACTH 250 µg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2011-08-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT02378298/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT02378298/SAP_001.pdf